CLINICAL TRIAL: NCT00575965
Title: Phase II Study of Simvastatin in Waldenstrom's Macroglobulinemia
Brief Title: Simvastatin in Waldenstrom's Macroglobulinemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual led to early study termination.
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Steven P. Treon, MD, PhD, Director, Bing Center, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-175
Record Dates: First submitted 2007-12-16; First posted 2007-12-18 (Estimated); Results first posted 2015-12-16 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-11

CONDITIONS: Waldenstrom's Macroglobulinemia
Keywords: simvastatin
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Simvastatin (Experimental): Simvastatin at 20 mg daily for the first week, then dose escalated weekly by 20 mg a day to a maximum of 80 mg daily by week 4. Patients were maintained on therapy until progression.
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Simvastatin — Oral tablets taken daily

SUMMARY:
This research study seeks to find new ways to treat people with Waldenstrom's Macroglobulinemia (WM). The study is for participants with slow growing WM who otherwise might not need therapy for at least 3-6 months. Simvastatin is a drug approved by the FDA for lowering cholesterol. In test tube studies the study drug appears to have direct anti-cancer effect against WM tumor cells and mast cells.

DETAILED DESCRIPTION:
OBJECTIVES:

To define objective response, time to progression and safety of Simvastatin in Waldenström's Macroglobulinemia.

STATISTICAL DESIGN:

For this phase II study, a single-stage design is used to evaluate the efficacy of Simvastatin. With a target enrollment of 30 participants, the 95% exact confidence bounds surrounding the response estimate will be no wider than +/- 19%.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Clinicopathological diagnosis of Waldenstrom's macroglobulinemia
* Measurable disease
* Slowly progressing disease not requiring therapy for at least 3-6 months and who do not meet consensus panel criteria for initiation of therapy
* ECOG Performance status of 0 or 1
* Adequate organ function as defined in the protocol
* Patients should agree to avoid grapefruit juice which is a major inhibitor of CYP 3A4

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study, or those who have not recovered from adverse events due to agents administered more than four weeks earlier
* Patients who have had rituximab within 3 months prior to entering the study
* Patients who have taken any Statin in the past
* Patients who take cyclosporin, danazol, or gemfibrozil will be excluded
* Prior history of rhabdomyolysis
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with the study requirements
* Pregnant or breastfeeding women
* HIV-positive
* Patients who take verapamil will be excluded
* Patients with active or history of liver disease
* Patients who consume more than three alcoholic beverages per day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Treon, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Outpatient Clinic at Dana Farber Cancer Institute
Pre-assignment Details: Patients with progressive nonsymptomatic disease on watch and wait were enrolled.
Groups:
- Simvastatin: Single arm, phase II study. All 18 patients received study drug.
Period: Overall Study
Arm/Group | Simvastatin
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Simvastatin
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Objective response is defined as achieving partial response or better on therapy based on the Consensus Panel Recommendations from the 2nd and 3rd International Workshop on WM [Weber et al, 2003; Kimby et al, 2005]. Complete Response (CR): Complete disappearance of serum monoclonal (SM) Immunoglobulin (Ig) E (IgE), measured centrally; resolution of adenopathy/organomegaly upon physical exam and computerized tomography (CT) scan; lymph nodes =<1.5 centimeters; absence of malignant cell by bone marrow histologic examination. Partial Response (PR): a >=50% reduction from baseline in the SM IgM concentration. Minor Response (MR): >=25%, but a <50% reduction of SM IgM from baseline.
Time Frame: Assessed at month 1 and 3 and thereafter every 3 months while on therapy. Median duration on treatment was 6 months (range 1-24 months).
Population: The analysis dataset is comprised of all evaluable patients. One patient was lost to follow-up within 3 weeks of enrollment and was unevaluable.
Measure: Number; unit: proportion of patients
Groups:
- Simvastatin: Simvastatin at 20 mg daily for the first week, then dose escalated weekly by 20 mg a day to a maximum of 80 mg daily by week 4. Patients were maintained on therapy until progression or up to 2 years.
Arm/Group | Simvastatin
Number analyzed (Participants) | 17
proportion of patients | 0.00

2. Primary Outcome: Progression-Free Survival
Description: Progression-free survival is the defined as the time from study entry to disease progression (PD) or death based on Kaplan-Meier estimates. Patients alibe without PD are censored at the date of last disease evaluation. PD is defined as a greater than 25% increase in serum IgM monoclonal protein levels from the lowest attained response value as determined by serum electrophoresis, confirmed by at least one other investigation, or progression of clinically significant disease related symptom(s). [Consensus panel criteria: Weber et al, 2003; Kimby et al, 2005].
Time Frame: Assessed at month 1 and 3 and thereafter every 3 months while on therapy; Assessed every 6 months for up to 2 years of follow-up. Median follow-up in this study cohort was 6 months (range 2-18 months).
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Simvastatin
Number analyzed (Participants) | 17
months | 6 [2.45 to 9.55]

ADVERSE EVENTS:
Time Frame: Assessed every 3 months on therapy up to day 30 post-therapy. Median duration on treatment was 6 months (range 1-24 months).
Description: The analysis dataset is comprised of all evaluable patients. One patient was lost to follow-up within 3 weeks of enrollment and was unevaluable.
Arm/Group | Simvastatin
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 4/17
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Simvastatin (N=17)
Elevated CPK (Musculoskeletal and connective tissue disorders) | 1 (1) — 1 grade 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3) — 3 patients with grade 2

LIMITATIONS AND CAVEATS:
Slow accrual led to early study termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No